CLINICAL TRIAL: NCT05400408
Title: Detection of Colorectal and Pancreatic Cancers Using Breath Analysis - Feasibility Study.
Brief Title: Chemical Profiling of Colorectal and Pancreatic Cancers Using Breath Analysis - Feasibility Study
Acronym: Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scentech Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRCPC-SMC-2021
Record Dates: First submitted 2022-05-24; First posted 2022-06-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer; Pancreatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Colorectal Cancer (Experimental): Subjects who were diagnosed as Colorectal Cancer patients by colonoscopy.
  Interventions: Diagnostic Test: VOX
- Pancreatic Cancer (Experimental): Subjects who were diagnosed as Pancreatic Cancer patients by Endoscopic Retrograde Cholangio Pancreatography.
  Interventions: Diagnostic Test: VOX
- Healthy volunteers (Other): Subjects who were found with no Colorectal or Pancreatic malignancies, by either colonoscopy or by Endoscopic Retrograde Cholangio Pancreatography.
  Interventions: Diagnostic Test: VOX

INTERVENTIONS:
Diagnostic Test: VOX — Breath Biopsy Analysis

SUMMARY:
Detection of Colorectal and Pancreatic Cancers Using Breath Analysis - Feasibility Study

DETAILED DESCRIPTION:
A diagnostic prospective study with no anticipated risks or constraints. Main Objective: To quantify differences in exhaled breath VOCs of patients with colorectal or pancreatic cancers compared with cohorts without cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85 years at the time of consent.
* Scheduled for colonoscopy or Endoscopic Retrograde Cholangio Pancreatography.
* Fasted >6 hours, consuming water only.
* Able to provide informed written consent.

Exclusion Criteria:

* Lacks capacity or is unable to provide informed written consent.
* Pregnant or lactating woman.
* Histologically confirmed cancer in any organ.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
identification of Volatile Organic Compounds that can be related to Colorectal malignancy. | Through the study completion, up to 1 year.
  Comparison of identity and concentration of Volatile Organic Compounds profile found among colorectal patients and the identity and concentration of Volatile Organic Compounds profile found among Healthy controls.

SECONDARY OUTCOMES:
Test Sensitivity and specificity for colorectal polyps. | Through the study completion, up to 1 year.
  Comparison of Volatile Organic Compounds found among subjects with and without colorectal polyps.
Test Sensitivity and specificity for pancreatic cancer. | Through the study completion, up to 1 year.
  Comparison of Volatile Organic Compounds found among pancreatic patients and Healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Haim Shirin, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Shamir Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No
No IPD is to be shared with other researchers.